CLINICAL TRIAL: NCT03808519
Title: Effects of n3 PUFA Supplementation on the Attenuation of Muscle Disuse Atrophy in Older Women
Brief Title: n3 PUFA and Muscle-disuse Atrophy in Older Women
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Stuart Phillips, Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: HiREB 1932
Record Dates: First submitted 2019-01-14; First posted 2019-01-17 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Muscle Atrophy; Muscle Disuse Atrophy; Sarcopenia
Keywords: n3 PUFA
MeSH Terms: conditions — Muscular Atrophy; Muscular Disorders, Atrophic; Sarcopenia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- n3 PUFA (Experimental): n3 PUFA (3000mg of Eicosapentaenoic acid per day and 1800mg of Docosahexaenoic acid per day)
  Interventions: Dietary Supplement: n3 PUFA-enriched fish oil
- Placebo (Placebo Comparator): Organic Sunflower Oil 5000mg per day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: n3 PUFA-enriched fish oil — 3000mg of Eicosapentaenoic acid per day and 1800mg of Docosahexaenoic acid per day
  Arms: n3 PUFA
Dietary Supplement: Placebo — Organic Sunflower Oil 5000mg per day
  Arms: Placebo

SUMMARY:
This study will examine the influence of n3 PUFA supplementation on the rate of muscle atrophy in older women undergoing 1 week of unilateral limb immobilization. Assessments in skeletal muscle strength and skeletal muscle volume will also me made before, after and in recovery from immobilization.

DETAILED DESCRIPTION:
Biological aging is associated with the loss of skeletal muscle mass and strength resulting in compromised metabolic function and mobility. Throughout life, individuals will also experience periods of reduced physical activity/muscle disuse that independently lower muscle mass and strength accelerating the aging process. More importantly, older adults (especially older women) that experience periods of muscle disuse are unable to recover muscle mass and strength. The losses in muscle mass with aging and disuse are underpinned by feeding-induced declines in rates of muscle protein synthesis. Thus, strategies to enhance muscle protein synthesis could have clinical implications for those who wish to maintain metabolic health and function during times of muscle disuse.

Supplementation with n3 PUFA-enriched fish oil has been shown to potentiate rates of muscle protein synthesis in response to simulated feeding in both younger and older adults. Fish oil supplementation also has been efficacious in enhancing skeletal muscle strength during a period of resistance exercise training. A previous study from our group demonstrated that younger women supplementing with n3 PUFA-enriched fish oil attenuated declines in skeletal muscle mass and strength during 2 weeks of immobilization. However, no study has examined the impact of fish oil supplementation to enhance muscle protein synthesis and offset declines in muscle mass/strength during a period of immobilization in older women.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Aged 55 - 75 years old
* non-smoking (for at least 2 years)
* > 5 years post-menopausal
* Body mass index (BMI) between 22 and 33 kg/m2
* Mini-Mental State Exam (MMSE) score > 20
* Acceptable medications include: Angiotensin Converting Enzyme (ACE), Beta-Blockers, Acetylsalicylic Acid, Calcium Channel blockers, Depression/Anxiety meds, Bisphosphonates (Fosamax®, Didrocal®, Actonel®, Aclasta®).

Exclusion Criteria:

* Any concurrent medical, orthopedic, or psychiatric condition that, in the opinion of the Investigators, would compromise the ability to comply with the study requirements.
* History of cancer within the last 5 years, except basal cell carcinoma, non-squamous skin carcinoma, prostate cancer, or carcinoma in situ with no significant progression over the past 2 years.
* Significant orthopedic, cardiovascular, pulmonary, renal, liver, infectious disease, immune disorder, or metabolic/endocrine disorders or other disease that would preclude oral n-3 PUFA supplement ingestion and/or assessment of safety and study objectives
* Current illnesses which could interfere with the study (e.g. prolonged severe diarrhea, regurgitation, difficulty swallowing)
* Participation in a study of an investigational product less than 60 days or 5 half-lives of the investigational product, whichever is longer, before enrollment in this study
* Hypersensitivity to the test product
* Excessive alcohol consumption (>21 units/week)
* Prior gastrointestinal bypass surgery
* History of bleeding diathesis, platelet or coagulation disorders, or antiplatelet/anticoagulation therapy
* Personal or family history of clotting disorder or deep vein thrombosis
* Concomitant use of corticosteroids, testosterone replacement therapy (ingestion, injection, or transdermal), or any anabolic steroid

Ages: 55 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — self- representation of gender identity
Enrollment: 8 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Muscle Cross-Sectional Area | Baseline (-28 days), pre-immobilization (0 days), post-immobilization (7 days), recovery (21 days)
  Changes in muscle cross-sectional area assessed by ultrasonography

SECONDARY OUTCOMES:
Integrated rates of muscle protein synthesis | pre-immobilization (0 days), post-immobilization (7 days), recovery (21 days)
  Change in muscle protein synthesis using doubly labelled water (D2O)
Skeletal muscle strength | Baseline (-28 days), pre-immobilization (0 days), post-immobilization (7 days), recovery (21 days)
  Change in skeletal muscle strength using the Biodex Dynamometer
Endothelial function | Baseline (-28 days), pre-immobilization (0 days), post-immobilization (7 days), recovery (21 days)
  Change in flow-mediated dilation
Vascular function | Baseline (-28 days), pre-immobilization (0 days), post-immobilization (7 days), recovery (21 days)
  Change in total femoral flow

CONTACTS AND LOCATIONS:
Overall Officials: Stuart M Phillips, PhD, Principal Investigator — McMaster University
Locations (1):
- Exercise Metabolism Research Laboratory, McMaster Univeristy, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No